CLINICAL TRIAL: NCT07131878
Title: Assesment of Treatment Outcomes of Aquired Aplastic Anemia in Children : A Retrospective and Prospective Cohort
Acronym: TTT
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abozaid, Resident doctor, Assiut University
Other Study IDs: Aquired Aplastic Anemia ttt
Record Dates: First submitted 2025-08-13; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Aplastic Anaemia (AA)
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- patient diagnosed with aplastic anemia from July 2023 to sept 2025
- patient diagnosed with aplastic anemia from Sept 2025 to July 2026

SUMMARY:
The goal of this observational study is to to assess of treatment Outcomes of Aquired Aplastic Anemia in children

DETAILED DESCRIPTION:
This study will be conducted to investigate the clinical outcomes, and treatment modalities of patients diagnosed with aquired aplastic anaemia at Assiut University children Hospital

The main question it aims to answer is:

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years diagnosed with acquired aplastic anemia, as confirmed by bone marrow examination and fulfilling diagnostic criteria (e.g., bone marrow cellularity <25% and at least two of the following: absolute neutrophil count <500/μL, platelet count <20,000/μL, absolute reticulocyte count <60,000/μL)123.
* The bone marrow biopsy should be compitable with diagnosis
* Diagnosed and/or treated at Assiut University Children's Hospital between Agust 2023 and Augst 2026.
* Patients with complete medical records, including diagnostic, laboratory, and treatment data

Exclusion Criteria:

* Patients with inherited bone marrow failure syndromes (e.g., Fanconi anemia, dyskeratosis congenita) as confirmed by genetic testing or family history21.
* Patients with incomplete or missing essential data in their medical records.
* Patients diagnosed outside the specified study period or managed primarily at other institutions.
* Patinets with neoplastic or granulomatous disease involving the bone marrow, systemic lupus erythematosus, AIDS, hypersplenism or other conditions associated with pancytopenia such as myelodysplastic syndrome,and paroxysmal nocturnal hemoglobinuria.
* Patients exposed to antineoplastic chemotherapy or radiotherapy were excluded

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged 1-18 years diagnosed with acquired aplastic anemia
Sampling Method: Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the treatment outcomes of children diagnosed with aplastic anemia. | July 2023-July 2026

SECONDARY OUTCOMES:
To assess response rates to various treatment modalities, including: oImmunosuppressive therapy (IST) oHematopoietic stem cell transplantation (HSCT) oSupportive care only | July 2023_July 2026

IPD SHARING:
Plan to Share IPD: No